CLINICAL TRIAL: NCT01031394
Title: Frequency of Aerobic/Resistance Training in Older Women
Acronym: SWEET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F050820002; R01AG027084 (NIH)
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Aging
Keywords: exercise; resistance training
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): 1 aerobic and 1 resistance training per week
  Interventions: Other: Frequency of Aerobic/Resistance Training - 3 to 3
- Group 2 (Active Comparator): 2 aerobic and 2 resistance training each per week
  Interventions: Other: Frequency of Aerobic/Resistance Training - 3 to 3
- Group 3 (Active Comparator): 3 aerobic and 3 resistance training per week
  Interventions: Other: Frequency of Aerobic/Resistance Training - 3 to 3

INTERVENTIONS:
Other: Frequency of Aerobic/Resistance Training - 3 to 3 — comparing group results based upon frequency of exercise
  Other Names: freqency of aerobic and resistance training

SUMMARY:
The objective of this study is to provide insight into the effects combined training frequency has on improving fitness, ease of physical activity, and maintenance of a high total energy expenditure. Such information is critical to our understanding of ways to improve well-being, quality of life, and independence of an aging population. 105 participants will be enrolled in this study. The length of time for your involvement in the study will be 32 weeks. You will undergo the procedures listed in this consent form on 3 separate occasions-initially at your entry, at 16 weeks and again at 32 weeks.

DETAILED DESCRIPTION:
Frequency of aerobic/resistance training in older women

Abstract Combined aerobic and resistance training have unique benefits for maintaining a physical activity (PA). However, the optimal training program for combining these two modes of training in older adults is unknown. This study builds on current and past studies showing that training induced gains in aerobic fitness, muscle strength, and ease of PA are important for maintaining an active lifestyle, a favorable body composition, and high bone density. Traditionally 3 d/wk combined training has been felt to be optimal while recent studies suggest 1 d/wk combined training may create similar adaptations as more frequent training. However, our previous and ongoing studies suggest that 1 d/wk combined aerobic and resistance training (C1) may be insufficient stimulus to induce optimal adaptations and that 3 d/wk combined training (C3) may be too frequent a stimulus for older adults. This study will enable us to compare the effects of C1, 2 d/wk combined training (C2), and C3 on fitness, body composition, ease of PA, PA, and total free-living energy expenditure (TEE). We hypothesize that C2 will result in a larger increase in muscle size, bone density, strength, aerobic capacity, power, ease of PA, PA, and TEE than either C1 or C3. Circulating cytokines and psychological mood states linked to chronic overstress will also be examined. Objectives: We will examine changes in circulating cytokines, mood states, muscle size, bone density, aerobic capacity, strength, power, ease of PA, PA, and TEE following 16 and 32 wks training. Design: We will to evaluate 78 (>60 yrs) Black and White women matched for age, race, and BMI into C1, C2, or C3 groups prior to, after 16, and after 32 wks training. Women will undergo evaluation of metabolic parameters in a General Clinical Research Center. Significance: This study should provide insight into the effects combined training frequency has on improving fitness, ease of PA, and maintenance of a high TEE. Such information is critical to our understanding of ways to improve well being, quality of life, and independence of an aging population.

ELIGIBILITY:
Inclusion Criteria:,

* healthy women over 60 years of age,
* Caucasian or African-American.

Exclusion Criteria:

* smoking,
* diabetes,
* osteoporosis,
* inability to coperform weight bearing exercises, currently performing to much exercise.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2004-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Use a repeated measures analysis to compare differences in TEE and other parameters among the 3 intervention groups across time | over 32 weeks of training

CONTACTS AND LOCATIONS:
Locations (1):
- UAB, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Martins C, Gower B, Hunter GR. Metabolic adaptation after combined resistance and aerobic exercise training in older women. Obesity (Silver Spring). 2022 Jul;30(7):1453-1461. doi: 10.1002/oby.23450. Epub 2022 Jun 21. PMID 35729736
- [Derived] Carter SJ, Baranauskas MN, Singh H, Martins C, Hunter GR. ARTE index revisited: linking biomarkers of cardiometabolic health with free-living physical activity in postmenopausal women. Am J Physiol Regul Integr Comp Physiol. 2022 Apr 1;322(4):R292-R298. doi: 10.1152/ajpregu.00075.2021. Epub 2022 Jan 26. PMID 35081314